CLINICAL TRIAL: NCT05925088
Title: Perspective of Patients With Chronic Pain in Evaluation of the Value of Online Exercise Videos
Brief Title: Exercise Videos - Perspectives of People Living With Chronic Pain
Status: Completed | Type: Observational
Sponsor: Walton Centre NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RG521-22
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Exercise
MeSH Terms: conditions — Chronic Pain; Motor Activity | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Focus group 1
  Interventions: Other: Focus group
- Focus group 2
  Interventions: Other: Focus group

INTERVENTIONS:
Other: Focus group — Participants will take part in a 1 hour focus group.

SUMMARY:
Exercise videos on the internet are used by millions worldwide to provide structure and motivation. They can guide exercise execution and play a role in helping people to maintain regular exercise.

On completion of the Pain Management Programme (PMP) at the Walton Centre, many patients are measurably more able bodied as a result (or at least part of a result) of regular engagement in exercise. Despite these positive outcomes and the patients stated intent to continue with exercise, many patients are struggling to maintain exercise in a meaningful way when re-assessed at their six month follow up appointment.

Patients have expressed that videos of the exercises would have motivated them to engage in sustained regular exercise in a more meaningful manner.

As physiotherapists, the investigators would like to ask a sample of patients on the PMP whether they anticipate exercise videos, reflecting the exercises practised on the PMP, would be beneficial for them to support maintenance/ sustainability of PMP exercises. Exercises practiced on the PMP include stretches, repeated movements in sitting, standing and lying, Pilates, yoga, normalised/functional movements and patients may like these exercises included in the videos.

The investigators plan to approach this using two focus groups followed by a qualitative analysis of recorded transcripts of the group discussions. Data would be analysed using a thematic analysis to establish key themes related to the research questions. The information gathered will inform the value of and content / format of specifically developed exercise videos.

The outcome of this project will inform the investigators of the use of exercise videos in this patient population and the value of this in encouraging people to keep up exercise over a sustained period. Other centres working with patients with chronic pain may be able to learn valuable lessons from this project in informing their own exercise promotion materials for their patients.

ELIGIBILITY:
Inclusion Criteria:

* Have attended a PMP at the Walton Centre within the last 12 months
* Aged 18+
* Able to provide written informed consent in English

Exclusion Criteria:

* Have not attended a PMP at the Walton Centre, or have attended >12 months ago

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain, who have attended a Pain Management Programme at the Walton Centre NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Themes related to focus group | 1-hour focus group
  Collection of qualitative data from focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Stevens, Principal Investigator — Physiotherapist
Locations (1):
- The Walton Centre NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided